CLINICAL TRIAL: NCT04206449
Title: Sleep Thermography for Diagnosis of Obstructive Sleep Apnea (OSA)
Brief Title: Sleep Thermography for Diagnosis of Obstructive Sleep Apnea (TERMOAPNEA)
Acronym: TERMOAPNEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Araba (Other)
Collaborators: Ibermática/i3B (Unknown); Instituto de Salud Carlos III (Other Government); Bioraba (Unknown)
Responsible Party: Principal Investigator, Carlos Javier Egea Santaolalla,Ph, Principal Investigator, MD, PhD, Hospital Universitario Araba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PI17/02011
Record Dates: First submitted 2019-11-06; First posted 2019-12-20 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: Infrared thermography system; Standard Polysomnography; Validity; Cost-effectiveness
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infrared thermography system (Experimental): Therapeutic decision taken with infrared thermography system, integrated in an expert diagnostic algorithm (TIS), to determine the sleep stages and Apnea-Hypopnea Index (AHI).
  Interventions: Other: Therapeutic decision Infrared thermgraphy system
- Standard Polysomnography (PSG) (Active Comparator): Therapeutic decision taken with Standard Polysomnography (PSG), to determine the sleep stages and Apnea-Hypopnea Index (AHI)
  Interventions: Other: Therapeutic decision PSG

INTERVENTIONS:
Other: Therapeutic decision PSG — Randomizing for therapeutic decision taken with Standard Polysomnography (PSG)
  Arms: Standard Polysomnography (PSG)
Other: Therapeutic decision Infrared thermgraphy system — Also randomizing for Infrared thermography system
  Arms: Infrared thermography system

SUMMARY:
To assess the diagnostic validity and cost-effectiveness of an infrared thermography system in adults with clinical suspicion of Obstructive Sleep Apnea (OSA).

DETAILED DESCRIPTION:
AIMS: To assess the diagnostic validity and cost-effectiveness of an infrared thermography system, integrated in an expert diagnostic algorithm (TIS), to determine the sleep stages and identify respiratory events, compared to conventional polysomnography (PSG) in adults with clinical suspicion of Obstructive Sleep Apnea (OSA).

METODOLOGY: DESIGN: Prospective, unicentric, randomized and blinded study carried out into two phases: Phase I: Development of the tool in 99 full valuable adults with suspected OSA (PSG recruitment, coordination and quality control, image capture, Information and development of the expert system); Phase II: Validation of the tool compared with the PSG in another group of 99 full valuable adults with suspected OSA. INSTRUMENTALIZATION: a) Clinical history and anthropometric variables; b) Sleep and quality of life questionnaires; c) PSG; d) TIS; e) Cost-effectiveness study.

ANALYSYS : The validity of the results of the TIS will be analyzed compared with the results of the PSG. The agreement measure will be established according to the different categories of the Apnea-Hypopnea Index (AHI), using ROC (Receiver Operating Characteristic) curves and the area under the curve. The investigators will also validate the therapeutic decisions made with PSG compared to those performed with the TIS. Finally, a cost-effectiveness study will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years to 75 years old, with clinical suspicion of OSA
* Written informed consent signed

Exclusion Criteria:

* Place of residence more than 100 km from the hospital
* Severe, unstable or exacerbated cardio-vascular, cerebro-vascular or respiratory disease, that makes it impossible to carry out adequate studies
* Presence of insomnia, depressive syndrome or epilepsia
* Patients diagnosed of any acute inflammatory episode of the cranium-maxillo-facial area or any systemic infection that develops with fever> 38 ºC at the time of testing
* Patient with malformation syndromes, Down syndrome and neuromuscular diseases
* Patient on active treatment with Positive continuous pressure (CPAP )

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | Baseline
  Count the respiratory events (apneas and hypopneas) that occur during sleep using a high sensitivity infrared thermal camera integrated in an expert diagnostic algorithm (TIS).

SECONDARY OUTCOMES:
Validation of the therapeutic decision | 6 month
  Analyze the concordance in the therapeutic decision using clinical findings and the results of Apnea-Hypopnea Index (AHI) from standard polysomnography (PSG) compared with data from infrared thermography system. In the Phase II.
Cost effectiveness analysis | 6 month
  Cost-efficacy evaluation: the analysis will be made in both arms based on intention to treat. Only direct costs will be analyzed: the cost of the use of polysomnography and infrared thermography system (Staff and consumable material).
Epworth Sleepiness Scale | baseline and at 6 month
  The Epworth Sleepiness Scale (the sum of 8 items score,0-3) can range from 0 to 24. Scores of 11-24 represent increasing levels of excessive daytime sleepiness.
STOP-Bang Questionnaire | baseline and at 6 month
  The questionnaire screens for obstructive sleep apnea (OSA):
  * Low risk of OSA: <3
  * High risk of OSA: ≥3
Berlin questionnaire | baseline and at 6 month
  The questionnaire consists of 3 categories related to the risk of having sleep apnea. Patients can be classified into High Risk or Low Risk based on their responses to the individual items and their overall scores in the symptom categories.
  * High Risk: if there are 2 or more categories where the score is positive.
  * Low Risk: if there is only 1 or no categories where the score is positive.
  Scoring Categories:
  * Category 1 is positive with 2 or more positive responses to questions 2-6
  * Category 2 is positive with 2 or more positive responses to questions 7-9
  * Category 3 is positive with 1 positive response and a BMI>30
Blood pressure | baseline and at 6 month
  Blood pressure measurements: systolic blood pressure and diastolic blood pressure
Anthropometric variables (Body mass index) | baseline and at 6 month
  Body mass index
Quality of life (EuroQOL test) | baseline and at 6 month
  Evaluate by EuroQOL test, is a standardised measure of health status. Description of the state of health in five dimensions (mobility, self-car, usual activities, pain/discomfort and anxiety/depression), each o wich is defined with three levels of severity, as measured by a Likert scale type (no problems, some problems and many problems or inability to activity).

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Duran-Cantolla, MD, Study Director — Hospital Universitario Araba
Locations (1):
- Hospital Universitario Araba, Vitoria-Gasteiz, Araba, Spain

REFERENCES:
- [Background] Durán-Cantolla J, Puertas FJ, Pin G y el Grupo Español de Sueño (GES).Documento de consenso nacional sobre el SAHS. Arch Bronconumol 2005;41(nº4):1-110.
- [Background] Lloberes P, Duran-Cantolla J, Martinez-Garcia MA, Marin JM, Ferrer A, Corral J, Masa JF, Parra O, Alonso-Alvarez ML, Teran-Santos J. Diagnosis and treatment of sleep apnea-hypopnea syndrome. Spanish Society of Pulmonology and Thoracic Surgery. Arch Bronconeumol. 2011 Mar;47(3):143-56. doi: 10.1016/j.arbres.2011.01.001. No abstract available. English, Spanish. PMID 21398016
- [Background] Duran J, Esnaola S, Rubio R, Iztueta A. Obstructive sleep apnea-hypopnea and related clinical features in a population-based sample of subjects aged 30 to 70 yr. Am J Respir Crit Care Med. 2001 Mar;163(3 Pt 1):685-9. doi: 10.1164/ajrccm.163.3.2005065. PMID 11254524
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Duran-Cantolla J, Mar J, de La Torre Munecas G, Rubio Aramendi R, Guerra L. [The availability in Spanish public hospitals of resources for diagnosing and treating sleep apnea-hypopnea syndrome]. Arch Bronconeumol. 2004 Jun;40(6):259-67. doi: 10.1016/s1579-2129(06)70096-9. Spanish. PMID 15161592
- [Background] Punjabi NM, Caffo BS, Goodwin JL, Gottlieb DJ, Newman AB, O'Connor GT, Rapoport DM, Redline S, Resnick HE, Robbins JA, Shahar E, Unruh ML, Samet JM. Sleep-disordered breathing and mortality: a prospective cohort study. PLoS Med. 2009 Aug;6(8):e1000132. doi: 10.1371/journal.pmed.1000132. Epub 2009 Aug 18. PMID 19688045
- [Background] Collop NA, Anderson WM, Boehlecke B, Claman D, Goldberg R, Gottlieb DJ, Hudgel D, Sateia M, Schwab R; Portable Monitoring Task Force of the American Academy of Sleep Medicine. Clinical guidelines for the use of unattended portable monitors in the diagnosis of obstructive sleep apnea in adult patients. Portable Monitoring Task Force of the American Academy of Sleep Medicine. J Clin Sleep Med. 2007 Dec 15;3(7):737-47. PMID 18198809
- [Background] Kushida CA, Littner MR, Morgenthaler T, Alessi CA, Bailey D, Coleman J Jr, Friedman L, Hirshkowitz M, Kapen S, Kramer M, Lee-Chiong T, Loube DL, Owens J, Pancer JP, Wise M. Practice parameters for the indications for polysomnography and related procedures: an update for 2005. Sleep. 2005 Apr;28(4):499-521. doi: 10.1093/sleep/28.4.499. PMID 16171294
- [Background] Mulgrew AT, Fox N, Ayas NT, Ryan CF. Diagnosis and initial management of obstructive sleep apnea without polysomnography: a randomized validation study. Ann Intern Med. 2007 Feb 6;146(3):157-66. doi: 10.7326/0003-4819-146-3-200702060-00004. PMID 17283346
- [Background] Epstein LJ, Kristo D, Strollo PJ Jr, Friedman N, Malhotra A, Patil SP, Ramar K, Rogers R, Schwab RJ, Weaver EM, Weinstein MD; Adult Obstructive Sleep Apnea Task Force of the American Academy of Sleep Medicine. Clinical guideline for the evaluation, management and long-term care of obstructive sleep apnea in adults. J Clin Sleep Med. 2009 Jun 15;5(3):263-76. PMID 19960649
- [Background] Van Someren EJ. More than a marker: interaction between the circadian regulation of temperature and sleep, age-related changes, and treatment possibilities. Chronobiol Int. 2000 May;17(3):313-54. doi: 10.1081/cbi-100101050. PMID 10841209
- [Background] Parmeggiani PL. Thermoregulation during sleep from the view point of homeostasis. Clinical Physiology of Sleep, American Physiological Society 1988, pp 159-69.
- [Background] van den Heuvel CJ, Noone JT, Lushington K, Dawson D. Changes in sleepiness and body temperature precede nocturnal sleep onset: evidence from a polysomnographic study in young men. J Sleep Res. 1998 Sep;7(3):159-66. doi: 10.1046/j.1365-2869.1998.00112.x. PMID 9785270
- [Background] Gilbert SS, van den Heuvel CJ, Ferguson SA, Dawson D. Thermoregulation as a sleep signalling system. Sleep Med Rev. 2004 Apr;8(2):81-93. doi: 10.1016/S1087-0792(03)00023-6. PMID 15033148
- [Background] Raymann RJ, Swaab DF, Van Someren EJ. Skin temperature and sleep-onset latency: changes with age and insomnia. Physiol Behav. 2007 Feb 28;90(2-3):257-66. doi: 10.1016/j.physbeh.2006.09.008. Epub 2006 Oct 27. PMID 17070562
- [Background] Parmeggiani PL, Agnati LF, Zamboni G, Cianci T. Hypothalamic temperature during the sleep cycle at different ambient temperatures. Electroencephalogr Clin Neurophysiol. 1975 Jun;38(6):589-96. doi: 10.1016/0013-4694(75)90159-5. PMID 50184
- [Background] Montgomery I, Trinder J, Paxton S, Harris D, Fraser G, Colrain I. Physical exercise and sleep: the effect of the age and sex of the subjects and type of exercise. Acta Physiol Scand Suppl. 1988;574:36-40. PMID 3245465
- [Background] Lack LC, Gradisar M, Van Someren EJ, Wright HR, Lushington K. The relationship between insomnia and body temperatures. Sleep Med Rev. 2008 Aug;12(4):307-17. doi: 10.1016/j.smrv.2008.02.003. PMID 18603220
- [Background] van den Heuvel CJ, Ferguson SA, Dawson D, Gilbert SS. Comparison of digital infrared thermal imaging (DITI) with contact thermometry: pilot data from a sleep research laboratory. Physiol Meas. 2003 Aug;24(3):717-25. doi: 10.1088/0967-3334/24/3/308. PMID 14509309